CLINICAL TRIAL: NCT05358028
Title: Comparison of Hand Arm Bimanual Intensive Technique With and Without Lower Extremity on Functional Status of Hemiplegic Cerebral Palsy
Brief Title: Effect of Hand Arm Bimanual Intensive Technique Including Lower Extremity (HABIT-IL) on Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ayesha Mahnoor
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hand arm bimanual intensive technique; Hemiplegic cerebral palsy; Functional status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand arm Bimanual intensive Technique including Lower extremity (HABIT-IL) (Experimental): Hand arm Bimanual activities involving Lower extremity
  Interventions: Other: Hand Arm Bimanual Intensive Technique including Lower Extremity (HABIT-IL)
- Hand Arm bimanual intensive Technique (HABIT) (Active Comparator): Hand arm Bimanual activities without involvement of lower extremity
  Interventions: Other: Hand Arm bimanual intensive Technique (HABIT)

INTERVENTIONS:
Other: Hand Arm Bimanual Intensive Technique including Lower Extremity (HABIT-IL) — HABIT-ILE along with the conventional Bobath treatment will be performed for 30 days in the form of groups for 3 hours, children will be performing individual activities.
  Functional task as maintaining ADL:
  i.Eating with spoon while standing ii. Combing hair while standing. iii. Counting cards while standing and putting them in box. Standing and walking I. standing with support of upper extremity II. walking with the help walkers III. walking on parallel bar playing activities: I. playing with cards while standings II. taking toys out of box and putting them in other box while standing III. grasping a fixed rod by hand and trying to maintain balance on physio stability ball
  Arms: Hand arm Bimanual intensive Technique including Lower extremity (HABIT-IL)
Other: Hand Arm bimanual intensive Technique (HABIT) — HAIBT along with the conventional Bobath treatment will be performed for 30 days in the form of groups for 3 hours, children will be performing individual activities HAIBT along with the conventional Bobth treatment will be performed for 30 days in the form of groups for 3 hours, children will be performing individual activities
  Playing activities on table:
  I. building towers with Lego blocks, II. Holding book by one hand and turning pages , III. Playing games with cards, IV. Drawing random impressions on paper, V. taking toys out of one box and placing them in other box one by one
  Activities of daily living :
  I. eating with spoon from bowel II. combing hair while sitting, III. opening of bottle cap for drinking water Age appropriate video games while sitting will be provided according to the ease of children
  Arms: Hand Arm bimanual intensive Technique (HABIT)

SUMMARY:
The aim of this study is to determine the functional status of upper extremity using HABIT & HABIT-ILE. And to compare the effects of HABIT with and without lower extremity technique on functional status of hemiplegic cerebral palsy

DETAILED DESCRIPTION:
Hemiplegic cerebral palsy children have impairments in bimanual coordination above and beyond their unilateral impairments .Hand-arm bimanual intensive therapy tends to show a constructive impact on hand function in children with hemi paretic cerebral palsy.

Hand-Arm Bimanual Intensive Therapy (HABIT) designed for children with unilateral CP, which when combines bimanual upper extremity training with activities involving the trunk and lower extremities making it HABIT-ILE.

A bimanual training program that continuously focusses on postural control and lower limb functional activity is all covered in HABIT-ILE Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) involves the concepts of motor skill learning and intensive training to both the UE and LE.

However it is not known that whether combined upper and lower extremity training in an intensive protocol is more efficacious or not thus Rationale of this study would be to figure out that if an intensive protocol is devised involving upper and lower extremities both would it be more product full or not. This study would be significant in a way that we know cerebral palsy is a lifelong challenging condition for both children and their caregivers thus new and emerging treatments can be fruitful for progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of hemiplegic cerebral palsy
* GMFCS level 2,3,4
* Ashworth scale 0-2

Exclusion Criteria:

* History of recent orthopedic surgery
* History of seizures
* Visual impairment

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
six minute walk test | 6 weeks
  The object of this test is to walk as far as possible for 6 minutes. the patient will walk back and forth in this hallway. Six minutes is a long time to walk, so the patient will be exerting. he will probably get out of breath or become exhausted. patients are permitted to slow down, to stop, and to rest as necessary. he may lean against the wall while resting, but resume walking as soon as patients are able. the patient will be walking back and forth around the cones. the patient should pivot briskly around the cones and continue back the other way without hesitation Predictive equation for males: 6 Minute Walk Distance (m) = 867 - (5.71 age, yrs) + (1.03 height, cm) Predictive equation for females: 6 Minute Walk Distance(m) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22 BMI).
Gross motor function measure | 6 week
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline.
  SCORING KEY 0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes NT = Not tested
Box And Block | 6 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke. The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. Clients are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Score each hand separately. Higher scores are indicative of better manual dexterity. During the performance of the BBT, the evaluator should be aware of whether the client's fingertips are crossing the partition. Blocks should be counted only when this condition is respected. Furthermore, if two blocks are transferred at once, only one block will be counted.
Assisting hand Assessment scale | 6 weeks
  AHA assesses the child's spontaneous and regular way of handling objects during play in natural settings, and is therefore a measure of usual everyday performance. AHA is appropriate to use for children with hemiplegic cerebral palsy (CP). 22 items consisting of observable actions, e.g. manipulates, varies grips, releases, and holds. The session is recorded and scored based on the 22 items on a 4-point rating scale evaluating quality of the performance (1=does not do, 4=effective).
  The range of sum scores is 22-88 points.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Mohi Ud Din Teaching Hospital (Mirpur AJK), Mirpur, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No